CLINICAL TRIAL: NCT01316159
Title: Prediction of Progression of Coronary Artery Disease and Clinical Outcome Using Vascular Profiling of Shear Stress and Wall Morphology
Brief Title: Prediction of Progression of Coronary Artery Disease (CAD) Using Vascular Profiling of Shear Stress and Wall Morphology
Acronym: PREDICTION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Shonan Kamakura General Hospital (Unknown); Cardiovascular Center Sakakibara Hospital (Unknown); Shiritsu Hakodate Hospital (Unknown); Sakurakai Takahashi Hospital (Unknown); Sapporo Higashi Tokushukai Hospital (Unknown); Kyoto Katsura Hospital (Unknown); Kokura Memorial Hospital (Other); Shonan Atsugi Hospital (Unknown); New Tokyo Hospital (Unknown); Aomori Prefectural Central Hospital (Unknown); Kanto Rosai Hospital (Unknown); Shin Koga Hospital (Unknown); Higashi Takarazuka Satoh Hospital (Unknown); Jichi Medical University (Other); Kumamoto Rosai Hospital (Unknown)
Responsible Party: Peter H. Stone, M.D., Study Chairman, Brigham & Women's Hospital, Harvard Medical School
Other Study IDs: PREDICTION
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Coronary Atherosclerosis; Acute Coronary Syndrome; Percutaneous Coronary Intervention; Endothelial Shear Stress; Arterial Remodeling
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although atherosclerosis is a systemic disease, its manifestations are focal and eccentric, and each coronary obstruction progresses, regresses, or remains quiescent in an independent manner. The focal and independent nature of atherosclerosis cannot be due solely to the presence of systemic risk factors such as hyperlipidemia, diabetes mellitus, cigarette smoking, and hypertension. Local factors that create a unique local environment are a major determinant of the behavior of atherosclerosis in a susceptible individual.

The vascular endothelium is in a unique and pivotal position to respond to the extremely dynamic forces acting on the vessel wall due to the complex 3-D geometry of the artery. Mechanical forces in general, and fluid shear stress (endothelial shear stress [ESS]) in particular, elicit a large number of humoral, metabolic and structural responses in endothelial cells.

Regions of disturbed flow, with low and oscillatory ESS (< 1.0 Pa), are intensely pro-atherogenic, pro-inflammatory, and pro-thrombotic, and correlate well with the localization of atherosclerotic lesions. These sites demonstrate intense accumulation of lipids, inflammatory cells, and matrix degrading enzymes which promote the formation of high-risk thin-cap fibroatheroma.

In contrast, physiologic laminar flow (1.0-2.5 Pa) is generally vasoprotective. However, as the obstruction progresses and further limits blood flow through a narrowed lumen, flow velocity and ESS may increase excessively (> 2.5 Pa) at the neck, and decrease abnormally at the outlet, increasing the likelihood of platelet activation and thrombus formation.

Identification of an early atherosclerotic plaque likely to progress and acquire characteristics leading to likelihood of rupture and, consequently, to precipitate an acute coronary event or rapid luminal obstruction, would permit more definitive pharmacologic or perhaps mechanical intervention prior to the occurrence of a cardiac event. The potential clinical value of identifying and "eradicating" plaques destined to become vulnerable before they actually become vulnerable is enormous.

The purpose of the PREDICTION Trial is to identify high-risk coronary lesions at an early time point in their evolution, to follow the natural history of these lesions over a 6-10 month period, and to confirm that these high-risk lesions are likely to rupture and cause an acute coronary syndrome (ACS) or develop rapid progression of a flow-limiting obstruction. The hypothesis is that local segments in the coronary arteries with low ESS and excessive expansive remodeling will be the sites where atherosclerotic plaque develops, progresses, and becomes high-risk, leading to a new cardiac event. This study is being conducted in Japan as patients are clinically evaluated with followup coronary angiography and IVUS in a routine manner at 6-10 months following their initial percutaneous coronary intervention (PCI) for an ACS.

This is a natural history and a clinical outcomes study in patients who initially present with an ACS. The natural history portion of the study is designed to describe the temporal progression of atherosclerosis in segments of coronary arteries with low ESS and expansive remodeling using intracoronary vascular profiling techniques utilizing intravascular ultrasound (IVUS) and coronary angiography. The clinical outcomes portion of the study is designed to evaluate the efficacy of coronary vascular profiling to predict segments of coronary arteries that will become areas of rapid plaque growth or rupture leading to recurrent major clinical coronary events.

Five hundred (500) patients with acute coronary syndrome undergoing PCI for a culprit lesion are to be enrolled in the study to undergo coronary vascular profiling at the time of the index catheterization procedure. Up to 374 consecutive patients with at least one low ESS subsegment are to have follow-up coronary angiography and IVUS at 6-10 months to allow for at least 300 patients with analyzable intracoronary vascular profiling data for assessment of lesion natural history. All patients are to have a one-year clinical follow-up to assess for new cardiac events, followed by two additional years of extended clinical followup.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Presentation with an ACS (unstable angina pectoris, non-ST elevation MI, or ST-elevation MI)
* Coronary artery disease with at least one coronary segment requiring percutaneous stent deployment using usual clinical indications
* At least 1 vessel suitable for IVUS not planned for PCI.
* Have the ability to understand the requirements of the study, provide written informed consent

Exclusion Criteria:

* Heart failure, defined as NYHA Class III or IV
* Unstable clinical status (ongoing anginal pain or hemodynamic or electrical instability)
* Left main disease or three vessel disease
* In the opinion of the investigator, significant coronary calcification precluding protocol evaluations
* Investigator determination of renal failure of sufficient severity such that additional contrast material is contraindicated
* Clinically significant valvular heart disease
* Investigator opinion of life expectancy < 12 months
* Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Studies requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational studies)
* Women who are pregnant, seeking to become pregnant or suspect they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease who present with an acute coronary syndrome and require cardiac catheterization and percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2007-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in coronary plaque thickness or area | From baseline to 6-10 month followup
  The primary endpoint is the change from baseline to 6-10 months in plaque thickness or area in the coronary segments identified to have low ESS at baseline.

SECONDARY OUTCOMES:
Change in other hemodynamic and morphology variables in segments with low ESS | 6-10 months
  Secondary endpoints will be changes from baseline to 6-10 months in the following coronary artery hemodynamic and morphology variables in segments with low ESS: change in lumen, change in EEM, change in ESS, change in arterial remodeling pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Antoniadis AP, Papafaklis MI, Takahashi S, Shishido K, Andreou I, Chatzizisis YS, Tsuda M, Mizuno S, Makita Y, Domei T, Ikemoto T, Coskun AU, Honye J, Nakamura S, Saito S, Edelman ER, Feldman CL, Stone PH. Arterial Remodeling and Endothelial Shear Stress Exhibit Significant Longitudinal Heterogeneity Along the Length of Coronary Plaques. JACC Cardiovasc Imaging. 2016 Aug;9(8):1007-9. doi: 10.1016/j.jcmg.2016.04.003. No abstract available. PMID 27491487
- [Derived] Stone PH, Saito S, Takahashi S, Makita Y, Nakamura S, Kawasaki T, Takahashi A, Katsuki T, Nakamura S, Namiki A, Hirohata A, Matsumura T, Yamazaki S, Yokoi H, Tanaka S, Otsuji S, Yoshimachi F, Honye J, Harwood D, Reitman M, Coskun AU, Papafaklis MI, Feldman CL; PREDICTION Investigators. Prediction of progression of coronary artery disease and clinical outcomes using vascular profiling of endothelial shear stress and arterial plaque characteristics: the PREDICTION Study. Circulation. 2012 Jul 10;126(2):172-81. doi: 10.1161/CIRCULATIONAHA.112.096438. Epub 2012 Jun 21. PMID 22723305